CLINICAL TRIAL: NCT06821243
Title: Multidimensional Assessment of Virus-associated Head and Neck Cancer Patients for the Discovery of Predictive Biomarkers to Guide Clinical Intervention
Brief Title: Patients with Human Papillomavirus-associated Head and Neck Cancer for the Discovery of Predictive Biomarkers to Guide Clinical Intervention
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: Università della Campania Luigi Vanvitelli (Unknown); Università di Napoli Federico II (Unknown); I.R.C.C.S. Fondazione Santa Lucia, Italy (Unknown)
Responsible Party: Sponsor
Other Study IDs: RS193/IRE/24
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Squamous Cell Carcinoma of Oropharynx
Keywords: carcinoma of the oropharynx; squamous cell carcinoma of the oropharynx; head and neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Oropharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — samples of tissue and liquid biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Prospective pilot study, non-interventional, of a biological/radiological nature, which involves the collection of tissue samples, and blood from patients suffering from squamous cell carcinoma of the oropharynx OPSCC for detection of HPV-DNA/RNA and immuno-phenotypic analysis of T cells, study of extracellular vesicles, and dosages of cytokines and chemokines involved in the immune response

DETAILED DESCRIPTION:
The study involves the collection of tissue samples, and blood from patients suffering from squamous cell carcinoma of the oropharynx OPSCC for detection of HPV-DNA/RNA and immuno-phenotypic analysis of T cells, study of extracellular vesicles, and dosages of cytokines and chemokines involved in the immune response. Radiological images will be collected during diagnosis, treatment and the care path, with exploratory and research purposes only, without the results modifying the care path and the diagnostic-therapeutic process of the patients participants. Molecular analyzes and/or material extraction will not be conducted genomic/protein of any kind. The objective is to observe the kinetics of the levels of HPV-DNA circulating in the blood patients with oropharynx cancers HPV related to the diagnosis and during the care pathway patient. The blood of HPV-negative patients will be tested to confirm that there are no copies of circulating HPV-DNA. The aim is to collect the information necessary to improve understanding and managing HPV-associated OPSCC.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell carcinomas of the oropharynx (OPSCC) candidates for surgical
* Age > 18 years
* ECOG performance status <_ 2
* Signature of informed consent (to participate in the study and data processing)

Exclusion Criteria:

* Presence of distant metastases at the time of diagnosis
* Previous head and neck cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by oropharynx squamous cell carcinoma (OPSCC) in head and neck district
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2026-07-24 (Estimated); Study Completion 2026-07-24 (Estimated)

PRIMARY OUTCOMES:
Observe the kinetics of HPV-DNA levels circulating in the blood | 24 months
  ctHPV DNA levels will be measured by digital PCR, 8 mL of blood will be collected in DNA BCT Streck tubes. The blood will be centrifuged a room temperature and frozen at -80°C until extraction. Total ctDNA will be extracted from 5 mL of plasma using the QIAamp Circulating Nucleic Acid Kit and will be quantified with a Qubit fluorometer. The ddPCR will be performed on a QX-200 platform and analyzed with QuantaSoft software v1.7.4.0917. Probes will be used for conserved regions of HPV E6 for HPV 16. Samples will be run with 5 cfDNA input to 10 ng and titered to optimize ddPCR performance, with a range of 1 to 20 ng of cfDNA total loaded per well. These reactions will be added to a DG8 cartridge along with 60mL of droplet generating oil. The drops will then be transferred to a plate from 96 wells and subjected to thermal cycles with the following conditions: 5 min at 95°C, 40 cycles at 94°C for 30 seconds, 55°C for 1 minute followed by 98°C for 10 min.

SECONDARY OUTCOMES:
Immuno-phenotyping at the tissue and blood level | 24 months
  Immuno-phenotyping at the tissue and blood level will be performed. Specific T cells for HPV will be identified by detecting the expression of the induced marker by activation (AIM) on the cell surface or by the production of intracellular cytokines, after exposure to HPV-derived peptide pools. AIM+ CD4+ T cells will be defined as positive for the expression of CD40L and CD69, while the expression of CD137 and CD69 will identify the subgroup CD8+ AIM+. The frequency and absolute number of specific CD4+ and CD8+ T cells will be determined HPV. Precise immunophenotyping will be performed using two panels antibodies. Innate immune cells and B lymphocytes will be investigated using a panel specific antibody to obtain a complete view of the patients' immune system
Isolation of extracellular vesicles | 24 months
  Extracellular vesicles will be isolated from patient plasma using Size exclusion chromatography to obtain homogeneous samples in terms of size using qEV35 columns, then stored in pre-filtered PBS at +4°C and used within 48 hours. Nanoparticle Tracking Analysis (NTA) will be used to determine the concentration and the size of vesicles isolated using Nanosight NS300. Membrane markers small EVs will be analyzed using the MACSPLex Human Exosomes kit (Milteny Biotec), for detection of 37 different membrane epitopes and two control isotypes.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS National Cancer Institute "Regina Elena", Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: No